CLINICAL TRIAL: NCT00527943
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of SCH 530348 in Addition to Standard of Care in Subjects With Acute Coronary Syndrome: Thrombin Receptor Antagonist for Clinical Event Reduction in Acute Coronary Syndrome (TRA•CER)
Brief Title: Trial to Assess the Effects of Vorapaxar (SCH 530348; MK-5348) in Preventing Heart Attack and Stroke in Particpants With Acute Coronary Syndrome (TRA•CER) (Study P04736)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The trial was terminated at the request of the Data and Safety Monitoring Board.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Duke Clinical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: P04736; TRA•CER; 2006-002809-31; MK-5348-014 (Other: Merck Study Number)
Record Dates: First submitted 2007-09-07; First posted 2007-09-11 (Estimated); Results first posted 2014-06-09 (Estimated); Last update posted 2018-09-21 (Actual); Status verified 2018-08

CONDITIONS: Atherosclerosis; Myocardial Ischemia; Myocardial Infarction
MeSH Terms: conditions — Atherosclerosis; Myocardial Ischemia; Myocardial Infarction | interventions — vorapaxar

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Loading oral dose of one 40 mg vorapaxar placebo tablet on Day 1, then one 2.5 mg vorapaxar placebo tablet daily, orally for at least 1 year in addition to current treatment of acute coronary syndrome, which will be continued to be administered as per current stand of care.
  Interventions: Drug: Placebo
- Vorapaxar (Experimental): Loading oral dose of one 40 mg vorapaxar tablet on Day 1, then one 2.5 mg vorapaxar tablet daily, orally for at least 1 year in addition to current treatment of acute coronary syndrome, which will be continued to be administered as per current stand of care.
  Interventions: Drug: Vorapaxar

INTERVENTIONS:
Drug: Vorapaxar — oral tablets; 40-mg loading dose on first day, followed by 2.5 mg once daily for at least 1 year
  Other Names: SCH 530348; MK-5348
  Arms: Vorapaxar
Drug: Placebo — oral tablets; matching placebo for vorapaxar; loading and maintenance dosing; once daily for at least 1 year
  Arms: Placebo

SUMMARY:
The study is designed to determine whether vorapaxar, when added to the existing standard of care (eg, aspirin, clopidogrel) for preventing heart attack and stroke in patients with acute coronary syndrome, will yield additional benefit over the existing standard of care in preventing heart attack and stroke.

The study is also designed to assess risk of bleeding with vorapaxar added to the standard of care versus the standard of care alone.

ELIGIBILITY:
Inclusion Criteria:

Men and women at least 18 years old with current clinical manifestation of non-ST-segment-elevation myocardial infarction (heart attack) according to the following three criteria:

* current symptoms of cardiac ischemia (chest pain leading to cardiac ischemia or heart attack)

AND

* either of the following:

  * concurrent elevation of troponin I or T, or of creatine kinase - myocardial band (CK-MB) to a level above the upper limit of normal, OR
  * concurrent appropriate electrocardiographic evidence

AND

* any one (or more) of the following:

  * age >= 55 years
  * documented history of prior heart attack or coronary revascularization (eg, angioplasty [PCI], coronary artery replacement [CABG])
  * diabetes (documented use of insulin or oral hypoglycemic[s])
  * documented history of peripheral arterial disease

Exclusion Criteria:

* history of intracranial hemorrhage or of central nervous system (CNS) surgery, tumor, or aneurysm
* any bleeding disorder or abnormality
* sustained severe hypertension or valvular heart disease
* current or recent platelet count <100,000 mm^3
* planned or ongoing treatment with a blood thinning medication
* pregnancy
* any significant medical or physiological condition or abnormality that could put the subject at increased risk or limit the subject's ability to participate for the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12944 (Actual)
Dates: Start 2007-12-01 (Actual); Primary Completion 2011-07-01 (Actual); Study Completion 2011-07-01 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Storey RF, Kotha J, Smyth SS, Moliterno DJ, Rorick TL, Moccetti T, Valgimigli M, Dery JP, Cornel JH, Thomas GS, Huber K, Harrington RA, Hord E, Judge HM, Chen E, Strony J, Mahaffey KW, Tricoci P, Becker RC, Jennings LK. Effects of vorapaxar on platelet reactivity and biomarker expression in non-ST-elevation acute coronary syndromes. The TRACER Pharmacodynamic Substudy. Thromb Haemost. 2014 May 5;111(5):883-91. doi: 10.1160/TH13-07-0624. Epub 2014 Jan 9. PMID 24402559
- [Result] Valgimigli M, Tricoci P, Huang Z, Aylward PE, Armstrong PW, Van de Werf F, Leonardi S, White HD, Widimsky P, Harrington RA, Cequier A, Chen E, Lokhnygina Y, Wallentin L, Strony J, Mahaffey KW, Moliterno DJ. Usefulness and safety of vorapaxar in patients with non-ST-segment elevation acute coronary syndrome undergoing percutaneous coronary intervention (from the TRACER Trial). Am J Cardiol. 2014 Sep 1;114(5):665-73. doi: 10.1016/j.amjcard.2014.05.054. Epub 2014 Jun 18. PMID 25129064
- [Derived] Batra G, Lindback J, Becker RC, Harrington RA, Held C, James SK, Kempf T, Lopes RD, Mahaffey KW, Steg PG, Storey RF, Swahn E, Wollert KC, Siegbahn A, Wallentin L. Biomarker-Based Prediction of Recurrent Ischemic Events in Patients With Acute Coronary Syndromes. J Am Coll Cardiol. 2022 Nov 1;80(18):1735-1747. doi: 10.1016/j.jacc.2022.08.767. PMID 36302586
- [Derived] Natale P, Palmer SC, Saglimbene VM, Ruospo M, Razavian M, Craig JC, Jardine MJ, Webster AC, Strippoli GF. Antiplatelet agents for chronic kidney disease. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD008834. doi: 10.1002/14651858.CD008834.pub4. PMID 35224730
- [Derived] Inohara T, Pieper K, Wojdyla DM, Patel MR, Jones WS, Tricoci P, Mahaffey KW, James SK, Alexander JH, Lopes RD, Wallentin L, Ohman EM, Roe MT, Vemulapalli S. Incidence, timing, and type of first and recurrent ischemic events in patients with and without peripheral artery disease after an acute coronary syndrome. Am Heart J. 2018 Jul;201:25-32. doi: 10.1016/j.ahj.2018.03.013. Epub 2018 Mar 28. PMID 29910052
- [Derived] Armaganijan LV, Alexander KP, Huang Z, Tricoci P, Held C, Van de Werf F, Armstrong PW, Aylward PE, White HD, Moliterno DJ, Wallentin L, Chen E, Harrington RA, Strony J, Mahaffey KW, Lopes RD. Effect of age on efficacy and safety of vorapaxar in patients with non-ST-segment elevation acute coronary syndrome: Insights from the Thrombin Receptor Antagonist for Clinical Event Reduction in Acute Coronary Syndrome (TRACER) trial. Am Heart J. 2016 Aug;178:176-84. doi: 10.1016/j.ahj.2016.05.012. Epub 2016 Jun 9. PMID 27502866
- [Derived] Popma CJ, Sheng S, Korjian S, Daaboul Y, Chi G, Tricoci P, Huang Z, Moliterno DJ, White HD, Van de Werf F, Harrington RA, Wallentin L, Held C, Armstrong PW, Aylward PE, Strony J, Mahaffey KW, Gibson CM. Lack of Concordance Between Local Investigators, Angiographic Core Laboratory, and Clinical Event Committee in the Assessment of Stent Thrombosis: Results From the TRACER Angiographic Substudy. Circ Cardiovasc Interv. 2016 May;9(5):e003114. doi: 10.1161/CIRCINTERVENTIONS.115.003114. PMID 27162212
- [Derived] Vranckx P, White HD, Huang Z, Mahaffey KW, Armstrong PW, Van de Werf F, Moliterno DJ, Wallentin L, Held C, Aylward PE, Cornel JH, Bode C, Huber K, Nicolau JC, Ruzyllo W, Harrington RA, Tricoci P. Validation of BARC Bleeding Criteria in Patients With Acute Coronary Syndromes: The TRACER Trial. J Am Coll Cardiol. 2016 May 10;67(18):2135-2144. doi: 10.1016/j.jacc.2016.02.056. PMID 27151345
- [Derived] Mahaffey KW, Hager R, Wojdyla D, White HD, Armstrong PW, Alexander JH, Tricoci P, Lopes RD, Ohman EM, Roe MT, Harrington RA, Wallentin L. Meta-analysis of intracranial hemorrhage in acute coronary syndromes: incidence, predictors, and clinical outcomes. J Am Heart Assoc. 2015 Jun 18;4(6):e001512. doi: 10.1161/JAHA.114.001512. PMID 26089177
- [Derived] Bagai A, Huang Z, Lokhnygina Y, Harrington RA, Armstrong PW, Strony J, White HD, Leonardi S, Held C, Van de Werf F, Wallentin L, Tricoci P, Mahaffey KW. Magnitude of troponin elevation and long-term clinical outcomes in acute coronary syndrome patients treated with and without revascularization. Circ Cardiovasc Interv. 2015 Jun;8(6):e002314. doi: 10.1161/CIRCINTERVENTIONS.115.002314. PMID 26025218
- [Derived] White HD, Huang Z, Tricoci P, Van de Werf F, Wallentin L, Lokhnygina Y, Moliterno DJ, Aylward PE, Mahaffey KW, Armstrong PW. Reduction in overall occurrences of ischemic events with vorapaxar: results from TRACER. J Am Heart Assoc. 2014 Jul 10;3(4):e001032. doi: 10.1161/JAHA.114.001032. PMID 25012288
- [Derived] Whellan DJ, Tricoci P, Chen E, Huang Z, Leibowitz D, Vranckx P, Marhefka GD, Held C, Nicolau JC, Storey RF, Ruzyllo W, Huber K, Sinnaeve P, Weiss AT, Dery JP, Moliterno DJ, Van de Werf F, Aylward PE, White HD, Armstrong PW, Wallentin L, Strony J, Harrington RA, Mahaffey KW. Vorapaxar in acute coronary syndrome patients undergoing coronary artery bypass graft surgery: subgroup analysis from the TRACER trial (Thrombin Receptor Antagonist for Clinical Event Reduction in Acute Coronary Syndrome). J Am Coll Cardiol. 2014 Mar 25;63(11):1048-57. doi: 10.1016/j.jacc.2013.10.048. Epub 2013 Nov 21. PMID 24211500
- [Derived] Tricoci P, Huang Z, Held C, Moliterno DJ, Armstrong PW, Van de Werf F, White HD, Aylward PE, Wallentin L, Chen E, Lokhnygina Y, Pei J, Leonardi S, Rorick TL, Kilian AM, Jennings LH, Ambrosio G, Bode C, Cequier A, Cornel JH, Diaz R, Erkan A, Huber K, Hudson MP, Jiang L, Jukema JW, Lewis BS, Lincoff AM, Montalescot G, Nicolau JC, Ogawa H, Pfisterer M, Prieto JC, Ruzyllo W, Sinnaeve PR, Storey RF, Valgimigli M, Whellan DJ, Widimsky P, Strony J, Harrington RA, Mahaffey KW; TRACER Investigators. Thrombin-receptor antagonist vorapaxar in acute coronary syndromes. N Engl J Med. 2012 Jan 5;366(1):20-33. doi: 10.1056/NEJMoa1109719. Epub 2011 Nov 13. PMID 22077816
- [Derived] TRA*CER Executive and Steering Committees. The Thrombin Receptor Antagonist for Clinical Event Reduction in Acute Coronary Syndrome (TRA*CER) trial: study design and rationale. Am Heart J. 2009 Sep;158(3):327-334.e4. doi: 10.1016/j.ahj.2009.07.001. PMID 19699853
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=P04736&kw=P04736&tab=access

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Prior to the planned study completion, the Data Safety Monitoring Board recommended that all participants stop treatment and that the study be closed-out. The protocol-defined target number of primary efficacy endpoints had been reached by this time. However, follow-up in the study was terminated earlier than planned.
Pre-assignment Details: The Intent to Treat (ITT) Population, defined as all enrolled participants who were randomly assigned to a treatment group.
Period: Overall Study
Arm/Group | Placebo | Vorapaxar
Started | 6471 | 6473
Received Treatment | 6441 | 6446
Completed | 6311 | 6327
Not Completed | 160 | 146

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vorapaxar | Total
Number analyzed (Participants) | 6471 | 6473 | 12944
Age, Customized [Number; unit: Participants]
  <65 years | 3369 | 3390 | 6759
  65 to <75 years | 2006 | 1973 | 3979
  >= 75 years | 1096 | 1110 | 2206
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1822 | 1810 | 3632
  Male | 4649 | 4663 | 9312

OUTCOME MEASURES:

1. Primary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Experienced Cardiovascular Death, Myocardial Infarction, Stroke, Recurrent Ischemia With Re-hospitalization, and/or Urgent Coronary Revascularization Within 2 Years From Randomization
Description: The time (in days) from study start to the first occurrence of any of the following clinical outcomes was recorded: cardiovascular (CV) death, myocardial infarction (MI), stroke, recurrent ischemia with re-hospitalization (RIR), and/or urgent coronary revascularization (UCR). A Clinical Endpoints Committee (CEC) reviewed and adjudicated each suspected efficacy endpoint event while blinded to treatment. Participants who did not have any endpoint event until last visit or participants who were lost to follow-up and had no event were censored at the time of last available information (last study visit). If a participant had a fatal event that was not part of a specific endpoint for analysis, they were censored at the time of death. The Kaplan-Meier estimate reports the percentage of participants who experienced at least 1 of the components of the primary composite efficacy endpoint within 2 years from randomization.
Time Frame: Up to 2 years
Population: Intent to Treat Population, defined as all participants who were randomly assigned to a treatment arm.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Vorapaxar
Number analyzed (Participants) | 6471 | 6473
Percentage of Participants | 19.9 | 18.5
Statistical Analysis 1: Comparison: Placebo vs Vorapaxar; Test type: Superiority or Other; p = 0.072, Cox Proportional Hazards Regression; Hazard Ratio calculated with covariates for treatment and stratification factors; Cox Proportional Hazard = 0.92, 95% CI 2-sided [0.85 to 1.01] — Hazard ratio calculated by dividing the Kaplan-Meier (KM) Estimate for vorapaxar by the KM Estimate for Placebo and correcting for covariates. A hazard ratio <1 would indicate a lower hazard associated with vorapaxar relative to placebo

2. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Experienced Cardiovascular Death, Myocardial Infarction, and/or Stroke Within 2 Years From Randomization
Description: The time (in days) from study start to the first occurrence of any of the following clinical outcomes was recorded: cardiovascular (CV) death, myocardial infarction (MI), and/or stroke. A CEC reviewed and adjudicated each suspected efficacy endpoint event while blinded to treatment. Participants who did not have any endpoint event until last visit or participants who were lost to follow-up and had no event were censored at the time of last available information (last study visit). If a participant had a fatal event that was not part of a specific endpoint for analysis, they were censored at the time of death. The Kaplan-Meier estimate reports the percentage of participants who experienced at least 1 of the components of the secondary composite efficacy endpoint within 2 years from randomization.
Time Frame: up to 2 years
Population: Intent to Treat Population, defined as all participants who were randomly assigned to a treatment arm.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Vorapaxar
Number analyzed (Participants) | 6471 | 6473
Percentage of Participants | 16.4 | 14.7
Statistical Analysis 1: Comparison: Placebo vs Vorapaxar; Test type: Superiority or Other; p = 0.018, Cox Proportional Hazards Regression; Hazard Ratio calculated with covariates for treatment and stratification factors; Cox Proportional Hazard = 0.89, 95% CI 2-sided [0.81 to 0.98] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Met Global Utilization of Streptokinase and Tissue Plasminogen Activator for Occluded Arteries (GUSTO) Moderate or Severe Bleeding Criteria Within 2 Years From Randomization
Description: Adverse events were categorized as "bleeding events" if the intensity of the event was other or more than would be normally expected in the given situation (eg, mild nosebleed in a person who does not normally have nosebleeds, greater bruising than expected for a given injury, greater volume of blood loss than expected for a given procedure). The investigator graded the intensity of bleeding events according to the GUSTO cooperative group criteria as follows: Mild , Moderate or Severe and the grading was adjudicated by the CEC. The Kaplan-Meier estimate reports the percentage of participants who experienced GUSTO moderate or severe bleeding within 2 years from randomization.
Time Frame: Up to 2 years
Population: As Treated Population, which included all participants who received at least 1 dose of study medication.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Vorapaxar
Number analyzed (Participants) | 6441 | 6446
Percentage of Participants | 5.8 | 7.6
Statistical Analysis 1: Comparison: Placebo vs Vorapaxar; Test type: Superiority or Other; p < 0.001, Cox Proportional Hazards Regression; Hazard Ratio calculated with covariates for treatment and stratification factors; Cox Proportional Hazard = 1.36, 95% CI 2-sided [1.18 to 1.57] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Experienced Clinically Significant Bleeding Within 2 Years From Randomization
Description: Adverse events were categorized as "bleeding events" if the intensity of the event was other or more than would be normally expected in the given situation (eg, mild nosebleed in a person who does not normally have nosebleeds, greater bruising than expected for a given injury, greater volume of blood loss than expected for a given procedure). The investigator graded the intensity of bleeding events according to the Thrombolysis in Myocardial Infarction (TIMI) Study Group criteria as major, minor or other. "Clinically Significant Bleeding" was defined as the composite of TIMI Major bleeding, TIMI Minor bleeding, or bleeding that required unplanned medical or surgical treatment or unplanned laboratory evaluation even if it did not meet the criteria for TIMI major or minor bleeding. The Kaplan-Meier estimate reports the percentage of participants who experienced clinically significant bleeding within 2 years from randomization.
Time Frame: Up to 2 years
Population: As Treated Population, which included all participants who received at least 1 dose of study medication.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Vorapaxar
Number analyzed (Participants) | 6441 | 6446
Percentage of Participants | 14.6 | 19.5
Statistical Analysis 1: Comparison: Placebo vs Vorapaxar; Test type: Superiority or Other; p < 0.001, Cox Proportional Hazards Regression; Hazard Ratio calculated with covariates for treatment and stratification factors; Cox Proportional Hazard = 1.41, 95% CI 2-sided [1.29 to 1.54] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Experienced CV Death, MI, Stroke, or UCR Within 2 Years From Randomization
Description: The time (in days) from study start to the first occurrence of any of the following clinical outcomes was recorded: CV death, MI, stroke, or UCR. A CEC reviewed and adjudicated each suspected efficacy endpoint event while blinded to treatment. Participants who did not have any endpoint event until last visit or participants who were lost to follow-up and had no event were censored at the time of last available information (last study visit). If a participant had a fatal event that was not part of a specific endpoint for analysis, they were censored at the time of death. The Kaplan-Meier estimate reports the percentage of participants who experienced CV death, MI, stroke, or UCR within 2 years from randomization.
Time Frame: Up to 2 years
Population: Intent to Treat Population, defined as all participants who were randomly assigned to a treatment arm.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Vorapaxar
Number analyzed (Participants) | 6471 | 6473
Percentage of Participants | 19.2 | 17.5
Statistical Analysis 1: Comparison: Placebo vs Vorapaxar; Test type: Superiority or Other; p = 0.038, Cox Proportional Hazards Regression; Hazard Ratio calculated with covariates for treatment and stratification factors; Cox Proportional Hazard = 0.91, 95% CI 2-sided [0.84 to 1.00] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Experienced CV Death or MI Within 2 Years From Randomization
Description: The time (in days) from study start to the first occurrence of any of the following clinical outcomes was recorded: CV death or MI. A CEC reviewed and adjudicated each suspected efficacy endpoint event while blinded to treatment. Participants who did not have any endpoint event until last visit or participants who were lost to follow-up and had no event were censored at the time of last available information (last study visit). If a participant had a fatal event that was not part of a specific endpoint for analysis, they were censored at the time of death. The Kaplan-Meier estimate reports the percentage of participants who experienced CV death or MI within 2 years from randomization.
Time Frame: Up to 2 years
Population: Intent to Treat Population, defined as all participants who were randomly assigned to a treatment arm.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Vorapaxar
Number analyzed (Participants) | 6471 | 6473
Percentage of Participants | 14.9 | 13.5
Statistical Analysis 1: Comparison: Placebo vs Vorapaxar; Test type: Superiority or Other; p = 0.027, Cox Proportional Hazards Regression; Hazard Ratio calculated with covariates for treatment and stratification factors; Cox Proportional Hazard = 0.90, 95% CI 2-sided [0.81 to 0.99] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Experienced All-cause Death, MI, Stroke, RIR, or UCR Within 2 Years From Randomization
Description: The time (in days) from study start to the first occurrence of any of the following clinical outcomes was recorded: all-cause death, MI, stroke, RIR, or UCR. A CEC reviewed and adjudicated each suspected efficacy endpoint event while blinded to treatment. Participants who did not have any endpoint event until last visit or participants who were lost to follow-up and had no event were censored at the time of last available information (last study visit). The Kaplan-Meier estimate reports the percentage of participants who experienced all-cause death, MI, stroke, RIR, or UCR within 2 years from randomization.
Time Frame: Up to 2 years
Population: Intent to Treat population, defined as all participants who were randomly assigned to a treatment arm.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Vorapaxar
Number analyzed (Participants) | 6471 | 6473
Percentage of Participants | 21.5 | 20.6
Statistical Analysis 1: Comparison: Placebo vs Vorapaxar; Test type: Superiority or Other; p = 0.174, Cox Proportional Hazards Regression; Hazard Ratio calculated with covariates for treatment and stratification factors; Cox Proportional Hazard = 0.94, 95% CI 2-sided [0.87 to 1.03] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Experienced All-cause Death, MI, Stroke, or UCR Within 2 Years From Randomization
Description: The time (in days) from study start to the first occurrence of any of the following clinical outcomes was recorded: all-cause death, MI, stroke, or UCR. A CEC reviewed and adjudicated each suspected efficacy endpoint event while blinded to treatment. Participants who did not have any endpoint event until last visit or participants who were lost to follow-up and had no event were censored at the time of last available information (last study visit). The Kaplan-Meier estimate reports the percentage of participants who experienced all-cause Death, MI, stroke, or UCR I within 2 years from randomization.
Time Frame: Up to 2 years
Population: Intent to Treat Population, defined as all participants who were randomly assigned to a treatment arm.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Vorapaxar
Number analyzed (Participants) | 6471 | 6473
Percentage of Participants | 20.8 | 19.6
Statistical Analysis 1: Comparison: Placebo vs Vorapaxar; Test type: Superiority or Other; p = 0.108, Cox Proportional Hazards Regression; Hazard Ratio calculated with covariates for treatment and stratification factors; Cox Proportional Hazard = 0.93, 95% CI 2-sided [0.86 to 1.02] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Experienced CV Death Within 2 Years From Randomization
Description: The time (in days) from study start to the CV death (if reported) was recorded. A CEC reviewed and adjudicated each suspected efficacy endpoint event while blinded to treatment. Participants who did not have any endpoint event until last visit or participants who were lost to follow-up and had no event were censored at the time of last available information (last study visit). If a participant had a fatal event that was not part of a specific endpoint for analysis, they were censored at the time of death. The Kaplan-Meier estimate reports the percentage of participants who experienced CV death within 2 years from randomization.
Time Frame: Up to 2 years
Population: Intent to Treat Population, defined as all participants who were randomly assigned to a treatment arm.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Vorapaxar
Number analyzed (Participants) | 6471 | 6473
Percentage of Participants | 3.8 | 3.8
Statistical Analysis 1: Comparison: Placebo vs Vorapaxar; Test type: Superiority or Other; p = 0.963, Cox Proportional Hazards Regression; Hazard Ratio calculated with covariates for treatment and stratification factors; Cox Proportional Hazard = 1.00, 95% CI 2-sided [0.83 to 1.22] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Experienced an MI Within 2 Years From Randomization
Description: The time (in days) from study start to the first occurrence of an MI was recorded. A CEC reviewed and adjudicated each suspected efficacy endpoint event while blinded to treatment. Participants who did not have any endpoint event until last visit or participants who were lost to follow-up and had no event were censored at the time of last available information (last study visit). If a participant had a fatal event that was not part of a specific endpoint for analysis, they were censored at the time of death. The Kaplan-Meier estimate reports the percentage of participants who experienced an MI within 2 years from randomization.
Time Frame: Up to 2 years
Population: Intent to Treat Population, defined as all participants who were randomly assigned to a treatment arm.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Vorapaxar
Number analyzed (Participants) | 6471 | 6473
Percentage of Participants | 12.5 | 11.1
Statistical Analysis 1: Comparison: Placebo vs Vorapaxar; Test type: Superiority or Other; p = 0.021, Cox Proportional Hazards Regression; Hazard Ratio calculated with covariates for treatment and stratification factors; Cox Proportional Hazard = 0.88, 95% CI 2-sided [0.79 to 0.98] — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Experienced RIR Within 2 Years From Randomization
Description: The time (in days) from study start to the first occurrence of RIR was recorded. A CEC reviewed and adjudicated each suspected efficacy endpoint event while blinded to treatment. Participants who did not have any endpoint event until last visit or participants who were lost to follow-up and had no event were censored at the time of last available information (last study visit). If a participant had a fatal event that was not part of a specific endpoint for analysis, they were censored at the time of death. The Kaplan-Meier estimate reports the percentage of participants who experienced RIR within 2 years from randomization.
Time Frame: Up to 2 years
Population: Intent to Treat Population, defined as all participants who were randomly assigned to a treatment arm
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Vorapaxar
Number analyzed (Participants) | 6471 | 6473
Percentage of Participants | 1.5 | 1.6
Statistical Analysis 1: Comparison: Placebo vs Vorapaxar; Test type: Superiority or Other; p = 0.418, Cox Proportional Hazards Regression; Hazard Ratio calculated with covariates for treatment and stratification factors; Cox Proportional Hazard = 1.14, 95% CI 2-sided [0.83 to 1.58] — [estimate comment as in outcome 1, analysis 1]

12. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Experienced UCR Within 2 Years From Randomization
Description: The time (in days) from study start to the first occurrence of UCR was recorded. A CEC reviewed and adjudicated each suspected efficacy endpoint event while blinded to treatment. Participants who did not have any endpoint event until last visit or participants who were lost to follow-up and had no event were censored at the time of last available information (last study visit). If a participant had a fatal event that was not part of a specific endpoint for analysis, they were censored at the time of death. The Kaplan-Meier estimate reports the percentage of participants who experienced UCR within 2 years from randomization.
Time Frame: Up to 2 years
Population: Intent to Treat Population, defined as all participants who were randomly assigned to a treatment arm.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Vorapaxar
Number analyzed (Participants) | 6471 | 6473
Percentage of Participants | 3.5 | 3.8
Statistical Analysis 1: Comparison: Placebo vs Vorapaxar; Test type: Superiority or Other; p = 0.493, Cox Proportional Hazards Regression; Hazard Ratio calculated with covariates for treatment and stratification factors; Cox Proportional Hazard = 1.07, 95% CI 2-sided [0.88 to 1.31] — [estimate comment as in outcome 1, analysis 1]

13. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Died From Any Cause Within 2 Years From Randomization
Description: The time (in days) from study start to death from any cause was recorded. A CEC reviewed and adjudicated each suspected efficacy endpoint event while blinded to treatment. Participants who did not have any endpoint event until last visit or participants who were lost to follow-up and had no event were censored at the time of last available information (last study visit). The Kaplan-Meier estimate reports the percentage of participants who died from any cause within 2 years from randomization.
Time Frame: Up to 2 years
Population: Intent to Treat Population, defined as all participants who were randomly assigned to a treatment arm.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Vorapaxar
Number analyzed (Participants) | 6471 | 6473
Percentage of Participants | 6.1 | 6.5
Statistical Analysis 1: Comparison: Placebo vs Vorapaxar; Test type: Superiority or Other; p = 0.515, Cox Proportional Hazards Regression; Hazard Ratio calculated with covariates for treatment and stratification factors; Cox Proportional Hazard = 1.05, 95% CI 2-sided [0.90 to 1.23] — [estimate comment as in outcome 1, analysis 1]

14. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Experienced a Stroke Within 2 Years From Randomization
Description: The time (in days) from study start to first experience of a stroke was recorded. A CEC reviewed and adjudicated each suspected efficacy endpoint event while blinded to treatment. Participants who did not have any endpoint event until last visit or participants who were lost to follow-up and had no event were censored at the time of last available information (last study visit). If a participant had a fatal event that was not part of a specific endpoint for analysis, they were censored at the time of death. The Kaplan-Meier estimate reports the percentage of participants who experienced a stroke within 2 years from randomization.
Time Frame: Up to 2 years
Population: Intent to Treat Population, defined as all participants who were randomly assigned to a treatment arm.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Vorapaxar
Number analyzed (Participants) | 6471 | 6473
Percentage of Participants | 2.1 | 1.9
Statistical Analysis 1: Comparison: Placebo vs Vorapaxar; Test type: Superiority or Other; p = 0.606, Cox Proportional Hazards Regression; Hazard Ratio calculated with covariates for treatment and stratification factors; Cox Proportional Hazard = 0.93, 95% CI 2-sided [0.70 to 1.23] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Description: Adverse events are reported using the As Treated Population, which included all participants who received at least 1 dose of study medication and are reported according to treatment received.
Arm/Group | Placebo | Vorapaxar
Serious Adverse Events (participants affected / at risk) | 1718/6441 | 1866/6446
Other Adverse Events (participants affected / at risk) | 832/6441 | 1081/6446
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=6441) | Vorapaxar (N=6446)
ANAEMIA (Blood and lymphatic system disorders) | 28 (29) | 55 (59)
COAGULOPATHY (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
EOSINOPHILIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
GRANULOCYTOPENIA (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
HAEMORRHAGIC ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
HAEMORRHAGIC DIATHESIS (Blood and lymphatic system disorders) | 1 (1) | 10 (10)
HEPARIN-INDUCED THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
HYPOCHROMIC ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 2 (3)
IDIOPATHIC THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 8 (8)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
LYMPHADENOPATHY MEDIASTINAL (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
MICROCYTIC ANAEMIA (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
NORMOCHROMIC NORMOCYTIC ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
SPLENIC INFARCTION (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
SPONTANEOUS HAEMATOMA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 34 (34) | 30 (30)
THROMBOCYTOSIS (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
ANGINA PECTORIS (Cardiac disorders) | 3 (3) | 6 (6)
ANGINA UNSTABLE (Cardiac disorders) | 0 (0) | 2 (2)
AORTIC VALVE DISEASE (Cardiac disorders) | 1 (1) | 0 (0)
AORTIC VALVE INCOMPETENCE (Cardiac disorders) | 0 (0) | 3 (3)
AORTIC VALVE STENOSIS (Cardiac disorders) | 1 (1) | 2 (2)
ARRHYTHMIA (Cardiac disorders) | 5 (5) | 6 (6)
ARRHYTHMIA SUPRAVENTRICULAR (Cardiac disorders) | 1 (1) | 3 (5)
ARTERIOSCLEROSIS CORONARY ARTERY (Cardiac disorders) | 0 (0) | 1 (1)
ARTERIOSPASM CORONARY (Cardiac disorders) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 93 (100) | 96 (113)
ATRIAL FLUTTER (Cardiac disorders) | 17 (17) | 17 (18)
ATRIAL RUPTURE (Cardiac disorders) | 1 (1) | 0 (0)
ATRIAL THROMBOSIS (Cardiac disorders) | 3 (3) | 0 (0)
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 1 (1) | 4 (4)
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 9 (9) | 9 (9)
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 6 (6) | 7 (7)
ATRIOVENTRICULAR DISSOCIATION (Cardiac disorders) | 1 (1) | 0 (0)
BIFASCICULAR BLOCK (Cardiac disorders) | 1 (1) | 0 (0)
BRADYARRHYTHMIA (Cardiac disorders) | 0 (0) | 1 (1)
BRADYCARDIA (Cardiac disorders) | 26 (26) | 14 (14)
BUNDLE BRANCH BLOCK LEFT (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 12 (12) | 9 (9)
CARDIAC ASTHMA (Cardiac disorders) | 2 (2) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 146 (191) | 142 (191)
CARDIAC FAILURE ACUTE (Cardiac disorders) | 1 (1) | 1 (1)
CARDIAC FAILURE CHRONIC (Cardiac disorders) | 4 (5) | 1 (1)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 35 (46) | 45 (53)
CARDIAC HYPERTROPHY (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC PERFORATION (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC TAMPONADE (Cardiac disorders) | 5 (5) | 4 (4)
CARDIAC VALVE DISEASE (Cardiac disorders) | 1 (1) | 0 (0)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 3 (3) | 2 (2)
CARDIOGENIC SHOCK (Cardiac disorders) | 39 (41) | 24 (24)
CARDIOMEGALY (Cardiac disorders) | 0 (0) | 1 (1)
CARDIOMYOPATHY (Cardiac disorders) | 4 (4) | 1 (1)
CARDIOPULMONARY FAILURE (Cardiac disorders) | 3 (3) | 3 (3)
CARDIOVASCULAR INSUFFICIENCY (Cardiac disorders) | 0 (0) | 1 (1)
CHORDAE TENDINAE RUPTURE (Cardiac disorders) | 0 (0) | 1 (1)
CONGESTIVE CARDIOMYOPATHY (Cardiac disorders) | 1 (1) | 0 (0)
COR PULMONALE (Cardiac disorders) | 0 (0) | 1 (1)
CORONARY ARTERY DISEASE (Cardiac disorders) | 6 (6) | 5 (5)
CORONARY ARTERY DISSECTION (Cardiac disorders) | 1 (1) | 1 (1)
CORONARY ARTERY INSUFFICIENCY (Cardiac disorders) | 0 (0) | 1 (1)
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 0 (0) | 1 (1)
DRESSLER'S SYNDROME (Cardiac disorders) | 1 (1) | 2 (2)
EXTRASYSTOLES (Cardiac disorders) | 1 (1) | 1 (1)
GASTROCARDIAC SYNDROME (Cardiac disorders) | 0 (0) | 1 (1)
HEART VALVE CALCIFICATION (Cardiac disorders) | 1 (1) | 0 (0)
INTRACARDIAC THROMBUS (Cardiac disorders) | 4 (4) | 2 (2)
ISCHAEMIC CARDIOMYOPATHY (Cardiac disorders) | 4 (4) | 2 (2)
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 1 (1) | 3 (3)
LEFT VENTRICULAR FAILURE (Cardiac disorders) | 0 (0) | 2 (3)
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 6 (6) | 5 (5)
MYOCARDIAL RUPTURE (Cardiac disorders) | 1 (1) | 1 (1)
MYOCARDITIS (Cardiac disorders) | 1 (1) | 0 (0)
MYOPERICARDITIS (Cardiac disorders) | 1 (1) | 0 (0)
NODAL ARRHYTHMIA (Cardiac disorders) | 2 (2) | 1 (1)
NODAL RHYTHM (Cardiac disorders) | 2 (2) | 0 (0)
PALPITATIONS (Cardiac disorders) | 6 (6) | 8 (8)
PAPILLARY MUSCLE RUPTURE (Cardiac disorders) | 1 (1) | 0 (0)
PERICARDIAL EFFUSION (Cardiac disorders) | 7 (7) | 7 (7)
PERICARDIAL HAEMORRHAGE (Cardiac disorders) | 8 (8) | 18 (19)
PERICARDITIS (Cardiac disorders) | 5 (5) | 3 (3)
PERICARDITIS CONSTRICTIVE (Cardiac disorders) | 1 (1) | 0 (0)
PLEUROPERICARDITIS (Cardiac disorders) | 1 (1) | 0 (0)
PRINZMETAL ANGINA (Cardiac disorders) | 0 (0) | 1 (1)
PULSELESS ELECTRICAL ACTIVITY (Cardiac disorders) | 2 (2) | 2 (2)
RESTRICTIVE CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 1 (2)
RIGHT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 1 (1) | 0 (0)
RIGHT VENTRICULAR FAILURE (Cardiac disorders) | 3 (3) | 0 (0)
SICK SINUS SYNDROME (Cardiac disorders) | 8 (8) | 7 (8)
SINOATRIAL BLOCK (Cardiac disorders) | 1 (1) | 1 (1)
SINUS ARREST (Cardiac disorders) | 0 (0) | 1 (1)
SINUS ARRHYTHMIA (Cardiac disorders) | 1 (1) | 1 (1)
SINUS BRADYCARDIA (Cardiac disorders) | 3 (3) | 3 (3)
SINUS TACHYCARDIA (Cardiac disorders) | 0 (0) | 2 (2)
STRESS CARDIOMYOPATHY (Cardiac disorders) | 1 (1) | 1 (1)
SUPRAVENTRICULAR TACHYARRHYTHMIA (Cardiac disorders) | 1 (1) | 0 (0)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 15 (15) | 9 (11)
TACHYCARDIA (Cardiac disorders) | 2 (2) | 2 (3)
TORSADE DE POINTES (Cardiac disorders) | 1 (1) | 1 (1)
TRICUSPID VALVE INCOMPETENCE (Cardiac disorders) | 1 (1) | 0 (0)
TRIFASCICULAR BLOCK (Cardiac disorders) | 1 (1) | 0 (0)
VENTRICLE RUPTURE (Cardiac disorders) | 0 (0) | 1 (1)
VENTRICULAR ARRHYTHMIA (Cardiac disorders) | 1 (1) | 3 (3)
VENTRICULAR DYSFUNCTION (Cardiac disorders) | 1 (1) | 0 (0)
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 1 (1) | 4 (4)
VENTRICULAR FIBRILLATION (Cardiac disorders) | 28 (33) | 30 (32)
VENTRICULAR TACHYARRHYTHMIA (Cardiac disorders) | 1 (1) | 0 (0)
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 36 (41) | 23 (29)
ARTERIOVENOUS MALFORMATION (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
ATRIAL SEPTAL DEFECT (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
GASTROINTESTINAL ANGIODYSPLASIA (Congenital, familial and genetic disorders) | 1 (1) | 2 (2)
GASTROINTESTINAL ANGIODYSPLASIA HAEMORRHAGIC (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL ARTERIOVENOUS MALFORMATION (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
HYDROCELE (Congenital, familial and genetic disorders) | 1 (1) | 1 (1)
PHIMOSIS (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
DEAFNESS (Ear and labyrinth disorders) | 1 (1) | 0 (0)
DEAFNESS NEUROSENSORY (Ear and labyrinth disorders) | 1 (1) | 0 (0)
EAR HAEMORRHAGE (Ear and labyrinth disorders) | 0 (0) | 1 (1)
SUDDEN HEARING LOSS (Ear and labyrinth disorders) | 1 (1) | 0 (0)
TINNITUS (Ear and labyrinth disorders) | 0 (0) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 10 (10) | 9 (9)
VERTIGO POSITIONAL (Ear and labyrinth disorders) | 3 (3) | 0 (0)
VESTIBULAR DISORDER (Ear and labyrinth disorders) | 0 (0) | 1 (1)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 1 (1) | 0 (0)
GOITRE (Endocrine disorders) | 0 (0) | 1 (1)
HYPERTHYROIDISM (Endocrine disorders) | 2 (2) | 0 (0)
HYPOTHYROIDISM (Endocrine disorders) | 1 (1) | 2 (2)
INAPPROPRIATE ANTIDIURETIC HORMONE SECRETION (Endocrine disorders) | 0 (0) | 1 (1)
TOXIC NODULAR GOITRE (Endocrine disorders) | 0 (0) | 1 (1)
ABNORMAL SENSATION IN EYE (Eye disorders) | 1 (1) | 0 (0)
CATARACT (Eye disorders) | 6 (7) | 4 (5)
CONJUNCTIVITIS (Eye disorders) | 0 (0) | 1 (1)
DIPLOPIA (Eye disorders) | 0 (0) | 1 (1)
EYE HAEMORRHAGE (Eye disorders) | 1 (1) | 0 (0)
GLAUCOMA (Eye disorders) | 2 (3) | 0 (0)
MACULAR HOLE (Eye disorders) | 0 (0) | 1 (1)
OPTIC ISCHAEMIC NEUROPATHY (Eye disorders) | 0 (0) | 1 (1)
RETINAL ARTERY OCCLUSION (Eye disorders) | 1 (1) | 2 (2)
RETINAL DETACHMENT (Eye disorders) | 1 (1) | 1 (1)
RETINAL VASCULAR THROMBOSIS (Eye disorders) | 1 (1) | 0 (0)
STRABISMUS (Eye disorders) | 1 (1) | 0 (0)
ULCERATIVE KERATITIS (Eye disorders) | 0 (0) | 1 (1)
VISUAL IMPAIRMENT (Eye disorders) | 1 (1) | 0 (0)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1 (1) | 0 (0)
ABDOMINAL HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 11 (15) | 11 (12)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 4 (4) | 9 (9)
ABDOMINAL STRANGULATED HERNIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
ABDOMINAL WALL HAEMATOMA (Gastrointestinal disorders) | 0 (0) | 1 (1)
ACUTE ABDOMEN (Gastrointestinal disorders) | 0 (0) | 1 (1)
ANAL FISTULA (Gastrointestinal disorders) | 1 (1) | 0 (0)
ANAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
ASCITES (Gastrointestinal disorders) | 2 (2) | 0 (0)
COELIAC DISEASE (Gastrointestinal disorders) | 1 (3) | 0 (0)
COLITIS (Gastrointestinal disorders) | 2 (2) | 1 (1)
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 5 (7) | 1 (1)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 1 (1) | 0 (0)
COLONIC POLYP (Gastrointestinal disorders) | 1 (1) | 2 (2)
CONSTIPATION (Gastrointestinal disorders) | 7 (9) | 6 (6)
CROHN'S DISEASE (Gastrointestinal disorders) | 1 (3) | 2 (2)
DIABETIC GASTROPARESIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 5 (6) | 8 (9)
DIARRHOEA HAEMORRHAGIC (Gastrointestinal disorders) | 0 (0) | 1 (1)
DIVERTICULAR PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
DIVERTICULUM (Gastrointestinal disorders) | 2 (2) | 1 (1)
DIVERTICULUM INTESTINAL (Gastrointestinal disorders) | 1 (1) | 0 (0)
DIVERTICULUM INTESTINAL HAEMORRHAGIC (Gastrointestinal disorders) | 0 (0) | 1 (1)
DUODENAL ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1)
DUODENAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 2 (2)
DUODENITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 2 (2)
DYSPHAGIA (Gastrointestinal disorders) | 1 (1) | 1 (1)
ENTERITIS (Gastrointestinal disorders) | 2 (2) | 0 (0)
ENTEROVESICAL FISTULA (Gastrointestinal disorders) | 0 (0) | 1 (1)
EROSIVE OESOPHAGITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
FAECALOMA (Gastrointestinal disorders) | 1 (1) | 2 (2)
FOOD POISONING (Gastrointestinal disorders) | 0 (0) | 2 (2)
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 4 (4) | 3 (4)
GASTRIC POLYPS (Gastrointestinal disorders) | 2 (2) | 0 (0)
GASTRIC ULCER (Gastrointestinal disorders) | 7 (8) | 7 (7)
GASTRIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 3 (3) | 2 (2)
GASTRIC ULCER PERFORATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTRIC VARICES HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 5 (6) | 14 (14)
GASTRITIS EROSIVE (Gastrointestinal disorders) | 3 (3) | 5 (5)
GASTRITIS HAEMORRHAGIC (Gastrointestinal disorders) | 1 (1) | 3 (3)
GASTRODUODENITIS (Gastrointestinal disorders) | 1 (1) | 1 (1)
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 1 (1) | 2 (2)
GASTROINTESTINAL EROSION (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 13 (13) | 26 (28)
GASTROINTESTINAL NECROSIS (Gastrointestinal disorders) | 0 (0) | 3 (3)
GASTROINTESTINAL PERFORATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROINTESTINAL ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 10 (10) | 7 (7)
GINGIVAL BLEEDING (Gastrointestinal disorders) | 0 (0) | 1 (1)
HAEMATEMESIS (Gastrointestinal disorders) | 10 (10) | 12 (12)
HAEMATOCHEZIA (Gastrointestinal disorders) | 5 (5) | 10 (10)
HAEMORRHAGIC EROSIVE GASTRITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 3 (3) | 4 (4)
HAEMORRHOIDS (Gastrointestinal disorders) | 3 (3) | 1 (1)
HYPERCHLORHYDRIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
ILEUS (Gastrointestinal disorders) | 3 (3) | 4 (4)
ILEUS PARALYTIC (Gastrointestinal disorders) | 1 (1) | 0 (0)
INGUINAL HERNIA (Gastrointestinal disorders) | 6 (6) | 16 (16)
INGUINAL HERNIA, OBSTRUCTIVE (Gastrointestinal disorders) | 0 (0) | 1 (1)
INTESTINAL HAEMATOMA (Gastrointestinal disorders) | 0 (0) | 1 (1)
INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 3 (3) | 5 (5)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 4 (4) | 4 (4)
INTESTINAL PERFORATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
LARGE INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
LARGE INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1)
LOCALISED INTRAABDOMINAL FLUID COLLECTION (Gastrointestinal disorders) | 0 (0) | 1 (1)
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 4 (4) | 3 (3)
MECHANICAL ILEUS (Gastrointestinal disorders) | 1 (1) | 0 (0)
MELAENA (Gastrointestinal disorders) | 26 (28) | 38 (40)
MESENTERIC VEIN THROMBOSIS (Gastrointestinal disorders) | 2 (2) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 3 (3) | 1 (1)
OESOPHAGEAL PERFORATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
OESOPHAGEAL STENOSIS (Gastrointestinal disorders) | 0 (0) | 2 (2)
OESOPHAGEAL ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0)
OESOPHAGEAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
OESOPHAGITIS (Gastrointestinal disorders) | 0 (0) | 5 (5)
OESOPHAGITIS HAEMORRHAGIC (Gastrointestinal disorders) | 1 (1) | 0 (0)
PANCREATIC CYST (Gastrointestinal disorders) | 1 (1) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 6 (6) | 10 (10)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 4 (4) | 4 (4)
PEPTIC ULCER (Gastrointestinal disorders) | 2 (2) | 3 (3)
PERIODONTITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
PERITONEAL HAEMATOMA (Gastrointestinal disorders) | 1 (1) | 0 (0)
PERITONITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
PHARYNGOESOPHAGEAL DIVERTICULUM (Gastrointestinal disorders) | 1 (1) | 0 (0)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 22 (22) | 26 (29)
REFLUX OESOPHAGITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
RETROPERITONEAL FIBROSIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
RETROPERITONEAL HAEMATOMA (Gastrointestinal disorders) | 1 (1) | 0 (0)
RETROPERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 6 (6) | 7 (7)
SMALL INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 5 (5) | 1 (1)
SUBILEUS (Gastrointestinal disorders) | 1 (1) | 0 (0)
TONGUE DISORDER (Gastrointestinal disorders) | 0 (0) | 1 (1)
TOOTHACHE (Gastrointestinal disorders) | 0 (0) | 1 (1)
UMBILICAL HERNIA (Gastrointestinal disorders) | 2 (2) | 1 (1)
UMBILICAL HERNIA, OBSTRUCTIVE (Gastrointestinal disorders) | 1 (1) | 0 (0)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 6 (7) | 10 (10)
VOMITING (Gastrointestinal disorders) | 8 (8) | 3 (3)
ASTHENIA (General disorders) | 3 (3) | 4 (4)
BLOODY DISCHARGE (General disorders) | 1 (1) | 0 (0)
CATHETER SITE HAEMATOMA (General disorders) | 16 (16) | 13 (13)
CATHETER SITE HAEMORRHAGE (General disorders) | 17 (17) | 23 (23)
CHEST DISCOMFORT (General disorders) | 5 (5) | 6 (6)
CHEST PAIN (General disorders) | 33 (42) | 29 (30)
CYST (General disorders) | 1 (1) | 0 (0)
DEVICE BREAKAGE (General disorders) | 2 (2) | 0 (0)
DEVICE DISLOCATION (General disorders) | 1 (1) | 2 (2)
DEVICE MALFUNCTION (General disorders) | 0 (0) | 2 (2)
DRUG INTOLERANCE (General disorders) | 1 (1) | 0 (0)
EXERCISE TOLERANCE DECREASED (General disorders) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 0 (0) | 3 (3)
GAIT DISTURBANCE (General disorders) | 1 (1) | 0 (0)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1 (1) | 1 (1)
GENERALISED OEDEMA (General disorders) | 1 (1) | 0 (0)
HERNIA (General disorders) | 0 (0) | 1 (1)
HERNIA OBSTRUCTIVE (General disorders) | 1 (1) | 1 (1)
HYPOTHERMIA (General disorders) | 0 (0) | 1 (1)
IMPAIRED HEALING (General disorders) | 1 (1) | 6 (6)
INFLAMMATION (General disorders) | 0 (0) | 1 (1)
INFLUENZA LIKE ILLNESS (General disorders) | 1 (1) | 0 (0)
INJECTION SITE HAEMORRHAGE (General disorders) | 1 (1) | 1 (1)
LOCAL SWELLING (General disorders) | 1 (1) | 0 (0)
MALAISE (General disorders) | 1 (1) | 0 (0)
MEDICAL DEVICE COMPLICATION (General disorders) | 1 (1) | 0 (0)
MUCOSAL INFLAMMATION (General disorders) | 1 (1) | 0 (0)
MULTI-ORGAN DISORDER (General disorders) | 2 (2) | 4 (4)
MULTI-ORGAN FAILURE (General disorders) | 11 (11) | 7 (7)
NECROSIS (General disorders) | 0 (0) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 112 (127) | 141 (158)
OEDEMA PERIPHERAL (General disorders) | 3 (3) | 4 (4)
PAIN (General disorders) | 1 (1) | 1 (1)
POLYP (General disorders) | 1 (1) | 0 (0)
PUNCTURE SITE REACTION (General disorders) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 6 (6) | 4 (4)
SECRETION DISCHARGE (General disorders) | 0 (0) | 1 (1)
SENSATION OF PRESSURE (General disorders) | 1 (1) | 0 (0)
SUDDEN CARDIAC DEATH (General disorders) | 1 (1) | 0 (0)
THROMBOSIS IN DEVICE (General disorders) | 1 (1) | 0 (0)
ULCER (General disorders) | 1 (1) | 0 (0)
ACUTE HEPATIC FAILURE (Hepatobiliary disorders) | 0 (0) | 1 (1)
BILE DUCT OBSTRUCTION (Hepatobiliary disorders) | 0 (0) | 1 (1)
BILE DUCT STONE (Hepatobiliary disorders) | 2 (2) | 4 (4)
BILIARY COLIC (Hepatobiliary disorders) | 2 (2) | 1 (1)
BILIARY DYSKINESIA (Hepatobiliary disorders) | 0 (0) | 1 (1)
CHOLANGITIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
CHOLANGITIS ACUTE (Hepatobiliary disorders) | 1 (1) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 18 (18) | 9 (9)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 10 (10) | 10 (10)
CHOLELITHIASIS (Hepatobiliary disorders) | 15 (15) | 13 (13)
GALLBLADDER DISORDER (Hepatobiliary disorders) | 1 (1) | 1 (1)
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
HEPATIC FAILURE (Hepatobiliary disorders) | 4 (4) | 2 (2)
HEPATIC STEATOSIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
HEPATITIS (Hepatobiliary disorders) | 0 (0) | 3 (3)
HEPATITIS ACUTE (Hepatobiliary disorders) | 2 (2) | 0 (0)
HEPATITIS TOXIC (Hepatobiliary disorders) | 0 (0) | 2 (2)
JAUNDICE (Hepatobiliary disorders) | 0 (0) | 1 (1)
LIVER DISORDER (Hepatobiliary disorders) | 1 (1) | 0 (0)
ALLERGY TO CHEMICALS (Immune system disorders) | 0 (0) | 1 (1)
AMYLOIDOSIS (Immune system disorders) | 0 (0) | 1 (1)
ANAPHYLACTIC REACTION (Immune system disorders) | 2 (2) | 1 (1)
ANAPHYLACTIC SHOCK (Immune system disorders) | 0 (0) | 1 (1)
ANTIPHOSPHOLIPID SYNDROME (Immune system disorders) | 1 (1) | 0 (0)
CONTRAST MEDIA ALLERGY (Immune system disorders) | 0 (0) | 1 (1)
DRUG HYPERSENSITIVITY (Immune system disorders) | 1 (1) | 1 (1)
HYPERSENSITIVITY (Immune system disorders) | 1 (1) | 3 (3)
SARCOIDOSIS (Immune system disorders) | 1 (1) | 0 (0)
ABDOMINAL ABSCESS (Infections and infestations) | 2 (2) | 3 (3)
ABDOMINAL INFECTION (Infections and infestations) | 1 (1) | 1 (1)
ABDOMINAL SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
ABSCESS LIMB (Infections and infestations) | 1 (1) | 0 (0)
ABSCESS ORAL (Infections and infestations) | 0 (0) | 1 (1)
ANAL ABSCESS (Infections and infestations) | 2 (3) | 4 (4)
APPENDICITIS (Infections and infestations) | 4 (4) | 9 (9)
APPENDICITIS PERFORATED (Infections and infestations) | 2 (2) | 0 (0)
ARTERIOVENOUS GRAFT SITE INFECTION (Infections and infestations) | 0 (0) | 1 (1)
ARTERITIS INFECTIVE (Infections and infestations) | 1 (1) | 0 (0)
ARTHRITIS INFECTIVE (Infections and infestations) | 2 (2) | 0 (0)
BACTERAEMIA (Infections and infestations) | 1 (1) | 2 (2)
BACTERIAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
BACTERIAL SEPSIS (Infections and infestations) | 1 (1) | 1 (1)
BORRELIA INFECTION (Infections and infestations) | 1 (1) | 1 (1)
BRONCHITIS (Infections and infestations) | 11 (12) | 18 (18)
BRONCHITIS VIRAL (Infections and infestations) | 0 (0) | 1 (1)
BRONCHOPNEUMONIA (Infections and infestations) | 4 (4) | 2 (2)
CELLULITIS (Infections and infestations) | 16 (16) | 25 (26)
CHEST WALL ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
CHOLECYSTITIS INFECTIVE (Infections and infestations) | 0 (0) | 1 (1)
CLOSTRIDIAL INFECTION (Infections and infestations) | 2 (2) | 0 (0)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 1 (1) | 0 (0)
CYSTITIS (Infections and infestations) | 2 (2) | 2 (2)
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 1 (1) | 0 (0)
DEVICE RELATED INFECTION (Infections and infestations) | 2 (2) | 0 (0)
DIABETIC FOOT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
DIVERTICULITIS (Infections and infestations) | 8 (9) | 13 (14)
ENDOCARDITIS (Infections and infestations) | 3 (3) | 2 (2)
ENTEROCOCCAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
ENTEROCOCCAL SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
ERYSIPELAS (Infections and infestations) | 5 (5) | 3 (4)
ESCHERICHIA SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
EYE INFECTION (Infections and infestations) | 0 (0) | 1 (1)
GANGRENE (Infections and infestations) | 4 (5) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 8 (9) | 12 (13)
GASTROENTERITIS NOROVIRUS (Infections and infestations) | 1 (1) | 0 (0)
GASTROENTERITIS SALMONELLA (Infections and infestations) | 0 (0) | 1 (1)
GASTROENTERITIS VIRAL (Infections and infestations) | 3 (3) | 4 (4)
GRAFT INFECTION (Infections and infestations) | 0 (0) | 2 (2)
GROIN ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
GROIN INFECTION (Infections and infestations) | 0 (0) | 1 (1)
H1N1 INFLUENZA (Infections and infestations) | 0 (0) | 1 (1)
HAEMATOMA INFECTION (Infections and infestations) | 2 (2) | 1 (1)
HEPATITIS B (Infections and infestations) | 0 (0) | 1 (1)
HEPATITIS C (Infections and infestations) | 0 (0) | 1 (1)
HERPES SIMPLEX (Infections and infestations) | 0 (0) | 1 (1)
HERPES ZOSTER (Infections and infestations) | 1 (1) | 3 (3)
HIV INFECTION (Infections and infestations) | 0 (0) | 1 (1)
IMPLANT SITE INFECTION (Infections and infestations) | 1 (1) | 0 (0)
INCISION SITE INFECTION (Infections and infestations) | 3 (3) | 2 (2)
INFECTED CYST (Infections and infestations) | 1 (1) | 0 (0)
INFECTED SEBACEOUS CYST (Infections and infestations) | 0 (0) | 1 (1)
INFECTED SKIN ULCER (Infections and infestations) | 0 (0) | 1 (1)
INFECTION (Infections and infestations) | 3 (3) | 0 (0)
INFECTIVE EXACERBATION OF CHRONIC OBSTRUCTIVE AIRWAYS DISEASE (Infections and infestations) | 1 (1) | 1 (2)
INFLUENZA (Infections and infestations) | 1 (1) | 2 (2)
INJECTION SITE ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
INTERVERTEBRAL DISCITIS (Infections and infestations) | 0 (0) | 1 (1)
KIDNEY INFECTION (Infections and infestations) | 0 (0) | 1 (1)
LEISHMANIASIS (Infections and infestations) | 0 (0) | 1 (1)
LEPROSY (Infections and infestations) | 0 (0) | 1 (1)
LIP INFECTION (Infections and infestations) | 0 (0) | 1 (1)
LOBAR PNEUMONIA (Infections and infestations) | 5 (5) | 6 (6)
LOCALISED INFECTION (Infections and infestations) | 1 (1) | 4 (4)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (3) | 3 (3)
LUNG INFECTION (Infections and infestations) | 6 (6) | 1 (1)
LUNG INFECTION PSEUDOMONAL (Infections and infestations) | 1 (1) | 0 (0)
LYMPH NODE ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
MEDIASTINITIS (Infections and infestations) | 4 (4) | 5 (5)
MENINGITIS ASEPTIC (Infections and infestations) | 0 (0) | 1 (1)
METAPNEUMOVIRUS INFECTION (Infections and infestations) | 0 (0) | 1 (1)
NECROTISING FASCIITIS (Infections and infestations) | 1 (1) | 0 (0)
NOCARDIOSIS (Infections and infestations) | 0 (0) | 1 (1)
ORCHITIS (Infections and infestations) | 1 (1) | 0 (0)
OSTEOMYELITIS (Infections and infestations) | 7 (7) | 6 (6)
OSTEOMYELITIS CHRONIC (Infections and infestations) | 1 (1) | 1 (1)
OTITIS MEDIA (Infections and infestations) | 1 (1) | 0 (0)
OTITIS MEDIA CHRONIC (Infections and infestations) | 1 (1) | 0 (0)
PELVIC ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
PERICARDITIS TUBERCULOUS (Infections and infestations) | 0 (0) | 1 (1)
PERIDIVERTICULAR ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
PERIRECTAL ABSCESS (Infections and infestations) | 2 (2) | 0 (0)
PERITONEAL ABSCESS (Infections and infestations) | 1 (1) | 1 (1)
PNEUMONIA (Infections and infestations) | 83 (93) | 100 (111)
PNEUMONIA BACTERIAL (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA HAEMOPHILUS (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA INFLUENZAL (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA KLEBSIELLA (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA PNEUMOCOCCAL (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA PRIMARY ATYPICAL (Infections and infestations) | 1 (1) | 0 (0)
POST PROCEDURAL INFECTION (Infections and infestations) | 3 (4) | 3 (3)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 6 (6) | 9 (9)
PSEUDOMEMBRANOUS COLITIS (Infections and infestations) | 0 (0) | 1 (2)
PSEUDOMONAS BRONCHITIS (Infections and infestations) | 0 (0) | 1 (1)
PSOAS ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
PYELONEPHRITIS (Infections and infestations) | 5 (5) | 1 (1)
PYOTHORAX (Infections and infestations) | 1 (1) | 1 (1)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 7 (7) | 4 (4)
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 1 (1) | 0 (0)
SCROTAL ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 23 (23) | 24 (25)
SEPTIC SHOCK (Infections and infestations) | 18 (18) | 11 (11)
SERRATIA INFECTION (Infections and infestations) | 1 (1) | 0 (0)
SHUNT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
SIALOADENITIS (Infections and infestations) | 1 (1) | 0 (0)
SINUSITIS (Infections and infestations) | 2 (2) | 0 (0)
SKIN INFECTION (Infections and infestations) | 1 (1) | 3 (3)
SMALL INTESTINE GANGRENE (Infections and infestations) | 1 (1) | 0 (0)
STAPHYLOCOCCAL ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 2 (2) | 3 (3)
STAPHYLOCOCCAL MEDIASTINITIS (Infections and infestations) | 1 (1) | 0 (0)
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
STERNITIS (Infections and infestations) | 0 (0) | 1 (1)
STITCH ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
STREPTOCOCCAL SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 6 (6) | 3 (3)
URINARY TRACT INFECTION (Infections and infestations) | 26 (27) | 23 (25)
UROSEPSIS (Infections and infestations) | 2 (2) | 8 (8)
VESTIBULAR NEURONITIS (Infections and infestations) | 1 (1) | 2 (2)
VIRAL INFECTION (Infections and infestations) | 3 (3) | 2 (2)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 0 (0)
WOUND INFECTION (Infections and infestations) | 12 (12) | 7 (7)
WOUND INFECTION STAPHYLOCOCCAL (Infections and infestations) | 1 (2) | 0 (0)
WOUND SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
ABDOMINAL INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ABDOMINAL WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ALCOHOL POISONING (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
ANAEMIA POSTOPERATIVE (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
ARTERIAL INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ARTERIOVENOUS FISTULA SITE HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
BACK INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
CARDIAC PROCEDURE COMPLICATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
CARDIAC VALVE RUPTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
CEREBRAL HAEMORRHAGE TRAUMATIC (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
COLLAPSE OF LUNG (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
COMMINUTED FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
CONCUSSION (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
CONFUSION POSTOPERATIVE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
CONTUSION (Injury, poisoning and procedural complications) | 1 (1) | 6 (8)
CRUSH INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
EXTRADURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
FACE INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
FALL (Injury, poisoning and procedural complications) | 16 (16) | 22 (22)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 4 (4) | 9 (9)
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
FOOT FRACTURE (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
FOREARM FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
GASTROINTESTINAL STOMA COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
GUN SHOT WOUND (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
HEAD INJURY (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
HEPATIC HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
HEPATIC RUPTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 5 (5) | 7 (7)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
INCISION SITE COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
INCISION SITE HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
INFLAMMATION OF WOUND (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
LACERATION (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
LIMB INJURY (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
LIMB TRAUMATIC AMPUTATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
MENISCUS LESION (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
MULTIPLE FRACTURES (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OPEN FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OPERATIVE HAEMORRHAGE (Injury, poisoning and procedural complications) | 11 (12) | 10 (10)
OVERDOSE (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
PATELLA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
PERIPROSTHETIC FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
POST PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 6 (6) | 3 (3)
POST PROCEDURAL DISCHARGE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
POST PROCEDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 91 (91) | 112 (114)
POSTOPERATIVE HERNIA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
POSTOPERATIVE ILEUS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
POSTOPERATIVE THORACIC PROCEDURE COMPLICATION (Injury, poisoning and procedural complications) | 5 (5) | 4 (4)
POSTOPERATIVE WOUND COMPLICATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
POSTPERICARDIOTOMY SYNDROME (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
PUBIS FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 2 (2) | 7 (8)
SHUNT MALFUNCTION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
SKULL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
SKULL FRACTURED BASE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SOFT TISSUE INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 2 (3)
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
SPLENIC RUPTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
STAB WOUND (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
STERNAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 2 (2) | 9 (9)
SUBDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
TENDON INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
TENDON RUPTURE (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
THERMAL BURN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 5 (5) | 0 (0)
TRANSPLANT FAILURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
TRAUMATIC LIVER INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
TRAUMATIC LUNG INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
URINARY RETENTION POSTOPERATIVE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
VASCULAR PROCEDURE COMPLICATION (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 5 (5) | 17 (17)
VASOPLEGIA SYNDROME (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
VENA CAVA INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
WOUND (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
WOUND COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
WOUND HAEMORRHAGE (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
WOUND SECRETION (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
WRIST FRACTURE (Injury, poisoning and procedural complications) | 6 (6) | 0 (0)
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Investigations) | 1 (1) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (1)
BLEEDING TIME PROLONGED (Investigations) | 1 (1) | 1 (1)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 1 (1) | 0 (0)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 1 (1)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 0 (0) | 1 (1)
BLOOD CREATINE PHOSPHOKINASE MB INCREASED (Investigations) | 0 (0) | 1 (1)
BLOOD CREATININE INCREASED (Investigations) | 1 (1) | 1 (1)
BLOOD CULTURE POSITIVE (Investigations) | 1 (1) | 0 (0)
BLOOD GLUCOSE ABNORMAL (Investigations) | 0 (0) | 1 (1)
BLOOD GLUCOSE INCREASED (Investigations) | 3 (3) | 1 (2)
BLOOD POTASSIUM DECREASED (Investigations) | 0 (0) | 1 (1)
BLOOD PRESSURE INCREASED (Investigations) | 0 (0) | 1 (1)
C-REACTIVE PROTEIN INCREASED (Investigations) | 1 (1) | 1 (1)
CARDIAC MONITORING ABNORMAL (Investigations) | 0 (0) | 1 (1)
CAROTID BRUIT (Investigations) | 0 (0) | 1 (1)
EJECTION FRACTION DECREASED (Investigations) | 3 (3) | 2 (2)
ELECTROCARDIOGRAM QRS COMPLEX PROLONGED (Investigations) | 1 (1) | 1 (1)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 3 (3) | 0 (0)
HAEMOGLOBIN DECREASED (Investigations) | 11 (11) | 12 (12)
HEART RATE IRREGULAR (Investigations) | 1 (1) | 0 (0)
HEPATIC ENZYME INCREASED (Investigations) | 4 (4) | 4 (4)
LIPOPROTEIN (A) INCREASED (Investigations) | 0 (0) | 1 (1)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 2 (2) | 1 (1)
OCCULT BLOOD POSITIVE (Investigations) | 0 (0) | 3 (3)
PLATELET COUNT DECREASED (Investigations) | 4 (5) | 4 (4)
TRANSAMINASES INCREASED (Investigations) | 0 (0) | 1 (1)
TROPONIN INCREASED (Investigations) | 1 (1) | 0 (0)
URINE OUTPUT DECREASED (Investigations) | 0 (0) | 1 (1)
WEIGHT DECREASED (Investigations) | 0 (0) | 2 (2)
WEIGHT INCREASED (Investigations) | 1 (1) | 0 (0)
CACHEXIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 10 (10) | 7 (9)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 11 (13) | 6 (6)
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 5 (5) | 9 (9)
DIABETIC FOOT (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 4 (4) | 3 (8)
ELECTROLYTE IMBALANCE (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
FLUID OVERLOAD (Metabolism and nutrition disorders) | 6 (7) | 2 (2)
FLUID RETENTION (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
GOUT (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 8 (8) | 7 (7)
HYPERGLYCAEMIC HYPEROSMOLAR NONKETOTIC SYNDROME (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 9 (10) | 5 (5)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 11 (11) | 10 (12)
HYPOGLYCAEMIC UNCONSCIOUSNESS (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 4 (4) | 4 (4)
IRON DEFICIENCY (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
LACTIC ACIDOSIS (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OBESITY (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (4)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5)
ARTHRITIS REACTIVE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
ARTICULAR CALCIFICATION (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 8 (8) | 8 (8)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BURSITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
CERVICAL SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
CHONDRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
COMPARTMENT SYNDROME (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
CRYSTAL ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
HAEMARTHROSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 9 (9) | 3 (3)
JOINT EFFUSION (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
KYPHOSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
MUSCLE HAEMORRHAGE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCLE TIGHTNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 19 (19) | 14 (16)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 5 (5) | 10 (10)
MYALGIA (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (6)
MYALGIA INTERCOSTAL (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MYOPATHY (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
MYOSCLEROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 22 (22) | 16 (16)
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 (3) | 4 (5)
POLYARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
SCOLIOSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
SPINAL COLUMN STENOSIS (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
SPINAL DISORDER (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
SPONDYLOLISTHESIS (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
SYMPATHETIC POSTERIOR CERVICAL SYNDROME (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
SYNOVIAL CYST (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
TENDONITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
TRIGGER FINGER (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ABDOMINAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
ADRENAL ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
ADRENAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 3 (3)
BENIGN LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BENIGN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BENIGN NEOPLASM OF BLADDER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BENIGN OESOPHAGEAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
BILE DUCT CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 9 (9)
BLADDER NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (5)
BLADDER TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
BRAIN NEOPLASM BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
BREAST NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BRONCHIAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
CARDIAC VALVE FIBROELASTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
CEREBRAL HAEMANGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
CHRONIC LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
CHRONIC MYELOMONOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
COLON ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (10) | 20 (20)
COLON CANCER STAGE II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
COLON CANCER STAGE III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
COLON NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
COLORECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
ENDOMETRIAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
ENDOMETRIAL CANCER STAGE I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
ENDOMETRIAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
FIBROMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 4 (4)
GASTRIC CANCER STAGE 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
GASTRIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
GASTROINTESTINAL CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
GASTROINTESTINAL TRACT ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
GASTROOESOPHAGEAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
HEPATIC NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
HODGKIN'S DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
HODGKIN'S DISEASE MIXED CELLULARITY STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
INTESTINAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
INTRAOCULAR MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
IRITIC MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
LARGE CELL CARCINOMA OF THE RESPIRATORY TRACT STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
LARYNGEAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
LIPOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
LUNG ADENOCARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
LUNG CARCINOMA CELL TYPE UNSPECIFIED STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4)
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 8 (8)
LUNG SQUAMOUS CELL CARCINOMA STAGE III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
MALIGNANT GLIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (4)
MEDIASTINUM NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
METASTASES TO BONE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
METASTASES TO LARYNX (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
METASTASES TO LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
METASTASES TO LUNG (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
METASTASES TO LYMPH NODES (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
METASTATIC MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
METASTATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
METASTATIC RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
METASTATIC SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
NASAL CAVITY CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
NEUROENDOCRINE CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
NON-SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
OESOPHAGEAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
OESOPHAGEAL CARCINOMA RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OVARIAN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
OVARIAN CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OVARIAN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
PAGET'S DISEASE OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PHAEOCHROMOCYTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0)
PITUITARY TUMOUR BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 7 (8)
PROSTATE CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
PROSTATE CANCER RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
PROSTATIC ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
RECTAL ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
RECTAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0)
RENAL CANCER RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
RENAL CELL CARCINOMA RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
RENAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
RENAL ONCOCYTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
SARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
SMALL CELL LUNG CANCER STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
SMALL INTESTINE CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
T-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
TESTIS CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
THYROID NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
TONGUE NEOPLASM MALIGNANT STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
UTERINE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
ALCOHOLIC SEIZURE (Nervous system disorders) | 1 (1) | 0 (0)
ATAXIA (Nervous system disorders) | 2 (2) | 1 (1)
BRACHIAL PLEXOPATHY (Nervous system disorders) | 0 (0) | 1 (1)
BRAIN MASS (Nervous system disorders) | 0 (0) | 1 (1)
BRAIN OEDEMA (Nervous system disorders) | 0 (0) | 1 (1)
CAROTID ARTERY DISEASE (Nervous system disorders) | 1 (1) | 2 (2)
CAROTID ARTERY OCCLUSION (Nervous system disorders) | 1 (1) | 1 (1)
CAROTID ARTERY STENOSIS (Nervous system disorders) | 11 (12) | 17 (18)
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 2 (2) | 0 (0)
CEREBELLAR HAEMORRHAGE (Nervous system disorders) | 1 (1) | 0 (0)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 (1) | 4 (4)
CEREBRAL HYPOPERFUSION (Nervous system disorders) | 0 (0) | 1 (1)
CERVICOBRACHIAL SYNDROME (Nervous system disorders) | 2 (2) | 1 (1)
CLUSTER HEADACHE (Nervous system disorders) | 1 (1) | 0 (0)
COMA (Nervous system disorders) | 1 (1) | 0 (0)
CONVULSION (Nervous system disorders) | 9 (9) | 6 (7)
CRANIAL NERVE PARALYSIS (Nervous system disorders) | 0 (0) | 1 (1)
CRITICAL ILLNESS POLYNEUROPATHY (Nervous system disorders) | 0 (0) | 1 (1)
DEMENTIA (Nervous system disorders) | 2 (2) | 1 (1)
DEMENTIA ALZHEIMER'S TYPE (Nervous system disorders) | 0 (0) | 1 (1)
DEMENTIA WITH LEWY BODIES (Nervous system disorders) | 0 (0) | 1 (1)
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 1 (1) | 0 (0)
DIABETIC NEUROPATHY (Nervous system disorders) | 1 (1) | 1 (1)
DIZZINESS (Nervous system disorders) | 10 (12) | 5 (5)
DYSAESTHESIA (Nervous system disorders) | 0 (0) | 1 (1)
DYSARTHRIA (Nervous system disorders) | 3 (3) | 0 (0)
ENCEPHALOPATHY (Nervous system disorders) | 4 (4) | 2 (2)
EPILEPSY (Nervous system disorders) | 4 (4) | 1 (1)
GRAND MAL CONVULSION (Nervous system disorders) | 2 (2) | 1 (2)
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 12 (13) | 33 (35)
HAEMORRHAGIC STROKE (Nervous system disorders) | 2 (2) | 0 (0)
HAEMORRHAGIC TRANSFORMATION STROKE (Nervous system disorders) | 0 (0) | 2 (2)
HEADACHE (Nervous system disorders) | 12 (12) | 2 (2)
HEMIPARESIS (Nervous system disorders) | 1 (1) | 1 (1)
HEPATIC ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 1 (1)
HYPERTENSIVE ENCEPHALOPATHY (Nervous system disorders) | 2 (2) | 0 (0)
HYPOAESTHESIA (Nervous system disorders) | 1 (1) | 0 (0)
HYPOKINESIA (Nervous system disorders) | 0 (0) | 1 (1)
HYPOTONIA (Nervous system disorders) | 0 (0) | 1 (1)
HYPOXIC-ISCHAEMIC ENCEPHALOPATHY (Nervous system disorders) | 1 (1) | 1 (1)
INTERCOSTAL NEURALGIA (Nervous system disorders) | 1 (1) | 0 (0)
INTRACRANIAL ANEURYSM (Nervous system disorders) | 1 (1) | 0 (0)
LETHARGY (Nervous system disorders) | 1 (1) | 1 (1)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 1 (1)
MENTAL IMPAIRMENT (Nervous system disorders) | 0 (0) | 1 (1)
MIGRAINE (Nervous system disorders) | 1 (1) | 0 (0)
MYASTHENIA GRAVIS (Nervous system disorders) | 1 (1) | 1 (1)
MYELOPATHY (Nervous system disorders) | 0 (0) | 1 (1)
NERVE COMPRESSION (Nervous system disorders) | 0 (0) | 2 (2)
NERVE DEGENERATION (Nervous system disorders) | 0 (0) | 1 (1)
NERVE ROOT COMPRESSION (Nervous system disorders) | 1 (1) | 0 (0)
NERVOUS SYSTEM DISORDER (Nervous system disorders) | 1 (1) | 0 (0)
NEURITIS (Nervous system disorders) | 1 (1) | 0 (0)
NEUROMYOPATHY (Nervous system disorders) | 1 (1) | 0 (0)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 2 (2) | 1 (1)
NORMAL PRESSURE HYDROCEPHALUS (Nervous system disorders) | 1 (1) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 5 (5) | 0 (0)
PARAPARESIS (Nervous system disorders) | 1 (1) | 0 (0)
PARKINSON'S DISEASE (Nervous system disorders) | 1 (1) | 1 (1)
PARTIAL SEIZURES (Nervous system disorders) | 0 (0) | 1 (1)
PERONEAL NERVE PALSY (Nervous system disorders) | 0 (0) | 1 (1)
PHRENIC NERVE PARALYSIS (Nervous system disorders) | 0 (0) | 1 (1)
PRESYNCOPE (Nervous system disorders) | 7 (7) | 4 (4)
PSYCHOMOTOR HYPERACTIVITY (Nervous system disorders) | 1 (1) | 0 (0)
SCIATICA (Nervous system disorders) | 3 (4) | 1 (1)
SEDATION (Nervous system disorders) | 1 (1) | 1 (1)
SENSORIMOTOR DISORDER (Nervous system disorders) | 1 (1) | 0 (0)
SENSORY LOSS (Nervous system disorders) | 0 (0) | 1 (1)
SPINAL CORD COMPRESSION (Nervous system disorders) | 1 (1) | 0 (0)
SPONDYLITIC MYELOPATHY (Nervous system disorders) | 0 (0) | 1 (1)
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 3 (3) | 3 (3)
SUBDURAL HYGROMA (Nervous system disorders) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 48 (48) | 44 (48)
SYRINGOMYELIA (Nervous system disorders) | 1 (2) | 0 (0)
TREMOR (Nervous system disorders) | 1 (1) | 0 (0)
VASCULAR ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 2 (2)
VERTEBRAL ARTERY STENOSIS (Nervous system disorders) | 0 (0) | 1 (1)
VIITH NERVE PARALYSIS (Nervous system disorders) | 1 (1) | 1 (1)
ABNORMAL BEHAVIOUR (Psychiatric disorders) | 1 (1) | 0 (0)
ADJUSTMENT DISORDER WITH MIXED DISTURBANCE OF EMOTION AND CONDUCT (Psychiatric disorders) | 0 (0) | 1 (1)
AGITATION (Psychiatric disorders) | 1 (1) | 0 (0)
ALCOHOL ABUSE (Psychiatric disorders) | 0 (0) | 1 (1)
ALCOHOL WITHDRAWAL SYNDROME (Psychiatric disorders) | 0 (0) | 2 (2)
ALCOHOLISM (Psychiatric disorders) | 1 (1) | 0 (0)
ANXIETY (Psychiatric disorders) | 7 (7) | 3 (3)
ANXIETY DISORDER (Psychiatric disorders) | 1 (1) | 0 (0)
BIPOLAR I DISORDER (Psychiatric disorders) | 1 (1) | 0 (0)
COMPLETED SUICIDE (Psychiatric disorders) | 2 (2) | 1 (1)
CONFUSIONAL STATE (Psychiatric disorders) | 4 (4) | 5 (5)
DELIRIUM (Psychiatric disorders) | 1 (1) | 2 (2)
DEPRESSION (Psychiatric disorders) | 8 (10) | 11 (15)
HALLUCINATION (Psychiatric disorders) | 1 (1) | 0 (0)
HALLUCINATION, VISUAL (Psychiatric disorders) | 1 (1) | 0 (0)
MAJOR DEPRESSION (Psychiatric disorders) | 2 (2) | 1 (2)
MENTAL STATUS CHANGES (Psychiatric disorders) | 3 (3) | 2 (2)
PANIC ATTACK (Psychiatric disorders) | 1 (1) | 0 (0)
PSYCHOTIC DISORDER (Psychiatric disorders) | 1 (1) | 1 (1)
SCHIZOAFFECTIVE DISORDER BIPOLAR TYPE (Psychiatric disorders) | 1 (1) | 0 (0)
SUBSTANCE ABUSE (Psychiatric disorders) | 0 (0) | 1 (1)
SUICIDAL IDEATION (Psychiatric disorders) | 2 (2) | 3 (3)
SUICIDE ATTEMPT (Psychiatric disorders) | 1 (1) | 3 (3)
TOBACCO WITHDRAWAL SYMPTOMS (Psychiatric disorders) | 0 (0) | 1 (1)
BLADDER DYSFUNCTION (Renal and urinary disorders) | 1 (1) | 0 (0)
CALCULUS BLADDER (Renal and urinary disorders) | 1 (1) | 1 (1)
CALCULUS URETERIC (Renal and urinary disorders) | 1 (1) | 4 (4)
CALCULUS URINARY (Renal and urinary disorders) | 2 (2) | 2 (2)
HAEMATURIA (Renal and urinary disorders) | 15 (16) | 31 (37)
HAEMORRHAGE URINARY TRACT (Renal and urinary disorders) | 2 (2) | 5 (6)
HYDRONEPHROSIS (Renal and urinary disorders) | 0 (0) | 1 (1)
NEPHROLITHIASIS (Renal and urinary disorders) | 6 (6) | 7 (7)
NEPHROPATHY (Renal and urinary disorders) | 1 (1) | 1 (1)
NEPHROPATHY TOXIC (Renal and urinary disorders) | 3 (3) | 1 (1)
NEPHROTIC SYNDROME (Renal and urinary disorders) | 1 (1) | 3 (3)
NEUROGENIC BLADDER (Renal and urinary disorders) | 1 (2) | 0 (0)
OBSTRUCTIVE UROPATHY (Renal and urinary disorders) | 0 (0) | 2 (2)
POLYURIA (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL ANEURYSM (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL ARTERY OCCLUSION (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL ARTERY STENOSIS (Renal and urinary disorders) | 3 (4) | 2 (2)
RENAL COLIC (Renal and urinary disorders) | 4 (5) | 6 (6)
RENAL CYST (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL DISORDER (Renal and urinary disorders) | 0 (0) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 50 (55) | 56 (61)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 36 (38) | 38 (39)
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 5 (5) | 8 (9)
RENAL IMPAIRMENT (Renal and urinary disorders) | 1 (1) | 2 (2)
RENAL MASS (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL TUBULAR NECROSIS (Renal and urinary disorders) | 1 (1) | 1 (1)
STRESS URINARY INCONTINENCE (Renal and urinary disorders) | 0 (0) | 1 (1)
TUBULOINTERSTITIAL NEPHRITIS (Renal and urinary disorders) | 0 (0) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 4 (4) | 6 (6)
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 1 (1)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 4 (4) | 9 (9)
BREAST INFLAMMATION (Reproductive system and breast disorders) | 1 (1) | 0 (0)
CYSTOCELE (Reproductive system and breast disorders) | 1 (1) | 0 (0)
EPIDIDYMITIS (Reproductive system and breast disorders) | 1 (1) | 1 (1)
GENITAL HAEMORRHAGE (Reproductive system and breast disorders) | 1 (1) | 1 (1)
OVARIAN CYST (Reproductive system and breast disorders) | 0 (0) | 1 (1)
PELVIC FLUID COLLECTION (Reproductive system and breast disorders) | 0 (0) | 1 (1)
POSTMENOPAUSAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 2 (2)
PROSTATITIS (Reproductive system and breast disorders) | 2 (2) | 2 (3)
PROSTATOMEGALY (Reproductive system and breast disorders) | 0 (0) | 1 (1)
RECTOCELE (Reproductive system and breast disorders) | 0 (0) | 1 (1)
UTERINE ENLARGEMENT (Reproductive system and breast disorders) | 0 (0) | 1 (1)
UTERINE PROLAPSE (Reproductive system and breast disorders) | 1 (1) | 0 (0)
VAGINAL PROLAPSE (Reproductive system and breast disorders) | 0 (0) | 1 (1)
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 14 (14)
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 16 (16) | 15 (16)
ALLERGIC GRANULOMATOUS ANGIITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ALVEOLITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
APNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 3 (3)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2)
BRONCHIAL HYPERREACTIVITY (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
BRONCHIAL OBSTRUCTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
BRONCHITIS CHRONIC (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 51 (71) | 44 (68)
CHYLOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
DIAPHRAGMATIC HERNIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DIAPHRAGMATIC PARALYSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 20 (20) | 20 (22)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
DYSPNOEA PAROXYSMAL NOCTURNAL (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 21 (22)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 7 (7)
HAEMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 3 (3)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HYDROTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
HYPERVENTILATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
LARYNGEAL OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
LARYNGEAL STENOSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
NASAL POLYPS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OBSTRUCTIVE AIRWAYS DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
OROPHARYNGEAL SWELLING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PHARYNGEAL HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 30 (31) | 32 (38)
PLEURAL HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 4 (4)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
PULMONARY ALVEOLAR HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
PULMONARY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 34 (34) | 20 (20)
PULMONARY EOSINOPHILIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
PULMONARY HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY MASS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 12 (13) | 19 (23)
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 26 (27) | 30 (30)
RESPIRATORY TRACT INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESTRICTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
TONSILLAR HYPERTROPHY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
VOCAL CORD POLYP (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DERMATITIS EXFOLIATIVE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DIABETIC ULCER (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
DYSHIDROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
NEUROPATHIC ULCER (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
PEMPHIGOID (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
PEMPHIGUS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
PSORIASIS (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
PURPURA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
SKIN HAEMORRHAGE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
SKIN LESION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
SKIN NECROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
STASIS DERMATITIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
SUBCUTANEOUS EMPHYSEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
URTICARIA (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
CARDIAC OPERATION (Surgical and medical procedures) | 2 (2) | 1 (1)
CATARACT OPERATION (Surgical and medical procedures) | 1 (1) | 1 (1)
DIABETES MELLITUS MANAGEMENT (Surgical and medical procedures) | 1 (1) | 0 (0)
WOUND DRAINAGE (Surgical and medical procedures) | 1 (1) | 0 (0)
ACCELERATED HYPERTENSION (Vascular disorders) | 2 (2) | 0 (0)
ANEURYSM (Vascular disorders) | 0 (0) | 1 (1)
AORTIC ANEURYSM (Vascular disorders) | 5 (5) | 6 (7)
AORTIC ANEURYSM RUPTURE (Vascular disorders) | 0 (0) | 1 (1)
AORTIC DISSECTION (Vascular disorders) | 6 (6) | 2 (2)
AORTIC DISSECTION RUPTURE (Vascular disorders) | 0 (0) | 1 (1)
AORTIC RUPTURE (Vascular disorders) | 1 (1) | 0 (0)
AORTIC STENOSIS (Vascular disorders) | 4 (4) | 4 (4)
AORTIC THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 4 (4) | 0 (0)
ARTERIAL STENOSIS LIMB (Vascular disorders) | 1 (1) | 0 (0)
ARTERIAL THROMBOSIS LIMB (Vascular disorders) | 0 (0) | 2 (3)
ARTERIOSCLEROSIS OBLITERANS (Vascular disorders) | 2 (2) | 1 (1)
ARTERIOVENOUS FISTULA (Vascular disorders) | 0 (0) | 1 (1)
CIRCULATORY COLLAPSE (Vascular disorders) | 2 (2) | 0 (0)
COELIAC ARTERY OCCLUSION (Vascular disorders) | 1 (1) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 10 (10) | 13 (13)
DIABETIC MACROANGIOPATHY (Vascular disorders) | 1 (1) | 0 (0)
EMBOLISM (Vascular disorders) | 1 (1) | 0 (0)
ESSENTIAL HYPERTENSION (Vascular disorders) | 2 (2) | 0 (0)
FEMORAL ARTERIAL STENOSIS (Vascular disorders) | 2 (2) | 1 (1)
FEMORAL ARTERY ANEURYSM (Vascular disorders) | 1 (1) | 0 (0)
FEMORAL ARTERY DISSECTION (Vascular disorders) | 0 (0) | 1 (1)
FEMORAL ARTERY OCCLUSION (Vascular disorders) | 3 (3) | 0 (0)
HAEMATOMA (Vascular disorders) | 7 (7) | 20 (26)
HAEMODYNAMIC INSTABILITY (Vascular disorders) | 2 (2) | 1 (1)
HAEMORRHAGE (Vascular disorders) | 12 (12) | 13 (13)
HYPERTENSION (Vascular disorders) | 23 (25) | 22 (24)
HYPERTENSIVE CRISIS (Vascular disorders) | 13 (13) | 20 (21)
HYPERTENSIVE EMERGENCY (Vascular disorders) | 2 (2) | 1 (1)
HYPOTENSION (Vascular disorders) | 28 (29) | 29 (29)
HYPOVOLAEMIC SHOCK (Vascular disorders) | 2 (2) | 0 (0)
ILIAC ARTERY STENOSIS (Vascular disorders) | 2 (2) | 3 (3)
INTERMITTENT CLAUDICATION (Vascular disorders) | 14 (16) | 9 (9)
INTRA-ABDOMINAL HAEMATOMA (Vascular disorders) | 0 (0) | 1 (1)
JUGULAR VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1)
LABILE HYPERTENSION (Vascular disorders) | 1 (1) | 0 (0)
LERICHE SYNDROME (Vascular disorders) | 1 (1) | 1 (1)
MALIGNANT HYPERTENSION (Vascular disorders) | 1 (1) | 0 (0)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 10 (10) | 6 (6)
PELVIC VENOUS THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 11 (12) | 13 (14)
PERIPHERAL ARTERY ANEURYSM (Vascular disorders) | 2 (2) | 0 (0)
PERIPHERAL ARTERY DISSECTION (Vascular disorders) | 0 (0) | 1 (1)
PERIPHERAL EMBOLISM (Vascular disorders) | 0 (0) | 1 (1)
PERIPHERAL ISCHAEMIA (Vascular disorders) | 9 (10) | 7 (7)
PERIPHERAL VASCULAR DISORDER (Vascular disorders) | 5 (7) | 8 (9)
PHLEBITIS (Vascular disorders) | 0 (0) | 2 (2)
POOR PERIPHERAL CIRCULATION (Vascular disorders) | 1 (1) | 0 (0)
SHOCK (Vascular disorders) | 1 (1) | 3 (3)
SHOCK HAEMORRHAGIC (Vascular disorders) | 0 (0) | 1 (1)
SUBCLAVIAN ARTERY STENOSIS (Vascular disorders) | 2 (2) | 1 (1)
SUBCLAVIAN STEAL SYNDROME (Vascular disorders) | 1 (1) | 0 (0)
TEMPORAL ARTERITIS (Vascular disorders) | 0 (0) | 1 (2)
THROMBOANGIITIS OBLITERANS (Vascular disorders) | 1 (1) | 0 (0)
THROMBOPHLEBITIS (Vascular disorders) | 0 (0) | 2 (2)
THROMBOPHLEBITIS SUPERFICIAL (Vascular disorders) | 1 (1) | 0 (0)
VARICOSE VEIN (Vascular disorders) | 0 (0) | 2 (2)
VASCULAR INSUFFICIENCY (Vascular disorders) | 0 (0) | 1 (1)
VASCULAR STENOSIS (Vascular disorders) | 1 (1) | 0 (0)
VASCULITIS (Vascular disorders) | 1 (1) | 0 (0)
VASODILATATION (Vascular disorders) | 0 (0) | 1 (1)
VENA CAVA THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
VENOUS THROMBOSIS (Vascular disorders) | 1 (1) | 1 (1)
VENOUS THROMBOSIS LIMB (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=6441) | Vorapaxar (N=6446)
HEADACHE (Nervous system disorders) | 385 (424) | 398 (451)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 228 (293) | 432 (552)
HYPERTENSION (Vascular disorders) | 310 (359) | 368 (399)

LIMITATIONS AND CAVEATS:
Prior to the planned study completion, the Data Safety Monitoring Board recommended that all participants stop treatment and that the study be closed-out. The protocol-defined target number of primary efficacy endpoints had been reached by this time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All draft publications will be submitted to the Publication Committee for review. Full-length papers will be submitted at least 45 days prior to submission to a journal. Abstracts or public presentations (eg, poster) will be submitted at least 14 days in advance.